CLINICAL TRIAL: NCT06297369
Title: Evaluation of the Effect of N-acetylcysteine in Preventing Cisplatin-Induced Toxicities in Cancer Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mahmoud Ibrahim, clinical pharmacist at ain shams university hospitals, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RHDIRB2020110301 REC #250
Record Dates: First submitted 2024-02-22; First posted 2024-03-07 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-02

CONDITIONS: Cisplatin Adverse Reaction; Cisplatin Nephrotoxicity; Cisplatin Induced Peripheral Neuropathy; Cancer Patients; Cisplatin Ototoxicity
Keywords: N-acetylcysteine; Ototoxicity; Cisplatin; Nephrotoxicity; Peripheral neuropathy
MeSH Terms: conditions — Ototoxicity; Peripheral Nervous System Diseases | interventions — Acetylcysteine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- control group (No Intervention): a. Group 1 (Control group, N = 30 patients) which will include patients who will receive cisplatin chemotherapy starting from 75mg/m2 for 4 cycles (21-28 days and or fractionated)
- treatment group (Active Comparator): b. Group 2 (N = 30 patients) will receive N-acetylcysteine 600 mg twice daily (Acetylcystein ® 600 mg effervescent instant granules sachets, Sedico, Egypt) with cisplatin chemotherapy for 4 cycles (21-28 days and or fractionated)
  Interventions: Drug: N acetyl cysteine

INTERVENTIONS:
Drug: N acetyl cysteine — N-acetylcysteine 600 mg twice daily (acetylcystein ® 600 mg effervescent instant granules sachets, Sedico, Egypt)
  Arms: treatment group

SUMMARY:
Evaluation of the Effect of N-acetylcysteine in Preventing Cisplatin-Induced Toxicities in Cancer Patients

DETAILED DESCRIPTION:
Cisplatin is a clinically advanced and highly effective anticancer drug used in the treatment of a wide variety of malignancies, Cisplatin was the first heavy metal compound to be used as an antineoplastic, and since its approval by the FDA in 1978, it is one of the most widely used agents in cancer therapy .

It has been used, sole or combined with other chemotherapeutic agents or even in combination with radiotherapy, in the treatment of several types of cancer, such as cancer of the testicles, ovarian, bladder, lung, head and neck, pancreas, breast, endometrium, esophagus, advanced cervical cancer, lymphomas, metastatic osteosarcomas and melanomas.

The therapeutic effect of cisplatin is significantly increased with dose-escalating, but high-dose therapy is limited by severe toxicities, with nephrotoxicity, neurotoxicity, and ototoxicity being the most important complications. In the case of nephrotoxicity, preventive measures such as saline hydration and osmotic diuresis are employed in clinical practice with minor success.

N-acetylcysteine (NAC) is a thiolic amino acid that has been reported to scavenge free radicals, replenish reduced glutathione (GSH), prevent its depletion, and inhibit lipid peroxidation (LPO). It can also restore the deterioration in the pro-oxidant/antioxidant balance via its metal-chelation activity.

Previous studies suggest that pre-administration of NAC attenuates carboplatin-induced injury in the cochlea of rats. As a GSH prodrug and antioxidant, NAC may ameliorate cochlear damage through a variety of mechanisms, such as providing a substrate for cochlear GSH synthesis, free radical scavenging, and inhibition of cell death pathway activation and necrosis.

To date, no clinical trial has been performed to evaluate the preventive potential of oral 1200 mg N-acetylcysteine on cisplatin-induced ototoxicity, hence this trial is designed to examine its effect on ototoxicity, nephrotoxicity, and neurotoxicity in cancer patients treated with cisplatin

Blood samples will be withdrawn from the study patients after enrollment to evaluate each of the following:

1. Complete blood picture (CBC) every cycle
2. Liver transaminases (AST and ALT) at baseline
3. Serum creatinine and blood urea nitrogen every cycle

Baseline glomerular filtration rate will be calculated according to the Cockcroft-Gault formula:

creatinine clearance (ml/min) = (140-age) x body weight plasma creatinine(mg/dl) x 72 The obtained value was multiplied by 0.85 for women.

* Baseline clinical investigations

  1. Audiometric test at baseline and every 2 cycles) patients will undergo conventional pure-tone audiometry in a soundproof room. The pure-tone thresholds for each ear will be measured at frequencies of 250, 500, 1000, 2000, 4000, and 8000 Hz).( bc cancer)
  2. Common terminology criteria for adverse event (CTCAE) version 4 (BC CANCER)
  3. The Functional Assessment of Cancer Therapy/Gynecologic Oncology Group-Neurotoxicity (FACT/GOG-Ntx) subscale.
* Follow-up and end-of-study evaluation The follow up of the patient will occur at the end of each cycle (after 21 days) and at the end of the study after receiving his or her 4th cycle.

ELIGIBILITY:
Inclusion Criteria:

* Patients are eligible for inclusion if they meet the following criteria:

  * Cancer patients aged >18 years receiving cisplatin-containing chemotherapy.
  * A cisplatin dose starting from 75 mg/m2.
  * Various cancer types.
  * Both males and females.
  * No history of organ transplantation or kidney dialysis.
  * Eastern cooperative oncology group performance (ECOG):0-2

Exclusion Criteria:

* Patients with peripheral neuropathy.
* Preexisting unilateral or bilateral moderate to severe sensorineural hearing loss
* Patients with speech discrimination affection or those who are unable to participate in audiologic evaluation
* Co-administration of ifosfamide with cisplatin, because of the known risk of nephrotoxicity.
* Pregnancy or lactation.
* Infection with the human immunodeficiency virus (HIV).
* Prior administration of cisplatin.
* Intraperitoneal chemotherapy.
* Inadequate liver function (bilirubin > 1.5 times upper normal limit [ULN] and alanine transaminase [ALT] or aspartate transaminase [AST] > 3 times the upper normal limit [ULN] or up to 5.0 upper normal limit [ULN] in the presence of hepatic metastases).
* Inadequate renal function (creatinine > 1.25 times upper normal limit [ULN], creatinine clearance < 50mL/min).
* Serious comorbid systemic disorder incompatible with the study (uncontrolled diabetes mellitus or hypertension, myocardial infarction within the last 6 months).
* Patients diagnosed with kidney cancer.
* Exposure to any nephrotoxic drugs or agents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
The occurrence of cisplatin-induced ototoxicity in the form of hearing loss. | 4 cycles of cisplatin (at base line and each cycle range from 21-28 days and or fractionated)
  hearing loss will be assessed using audiometry

SECONDARY OUTCOMES:
The occurrence of cisplatin-induced nephrotoxicity. | 4 cycles of cisplatin (at base line and each cycle range from 21-28 days and or fractionated)
  nephrotoxicity will be assessed using serum creatinine and blood urea nitrogen.
The occurrence of cisplatin-induced peripheral neuropathy. | 4 cycles of cisplatin (at base line and each cycle range from 21-28 days and or fractionated)
  peripheral neuropathy will be assessed using Common terminology criteria for adverse event (CTCAE)
The occurrence of cisplatin-induced peripheral neuropathy. | 4 cycles of cisplatin (at base line and each cycle range from 21-28 days and or fractionated)
  peripheral neuropathy will be assessed using The Functional Assessment of Cancer Therapy/Gynecologic Oncology Group-Neurotoxicity (FACT/GOG-Ntx) subscale
The occurrence of cisplatin-induced peripheral neuropathy. | 4 cycles of cisplatin (at base line and each cycle range from 21-28 days and or fractionated)
  peripheral neuropathy will be assessed using DouleurNeuropathique 4 Questions ( dn4 questionnaire)

CONTACTS AND LOCATIONS:
Overall Officials: mahmoud ibrahim, Principal Investigator — Ain Shams University
Locations (1):
- Department of Clinical Oncology and Nuclear Medicine, Ain Shams University Hospitals, Cairo, Egypt., Cairo, Egypt